CLINICAL TRIAL: NCT02727179
Title: Prospective and Randomized Study Comparing Open vs Laparoscopic Liver Surgery for Colorectal Liver Metastases
Brief Title: Open vs Laparoscopic Liver Surgery for Colorectal Liver Metastases
Acronym: LapOpHuva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Ricardo Robles Campos, MD, PHD, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUVA-0515
Record Dates: First submitted 2016-03-14; First posted 2016-04-04 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Liver Metastasis; Laparoscopic Liver Resection
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic group (Experimental): Liver resection performed by laparoscopic approach
  Interventions: Procedure: Liver resection
- Open group (Active Comparator): Liver resection performed by open approach
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — The investigators perform an anatomical liver resections or wedge resections depending on tumour's location and tumour's characteristics

SUMMARY:
This study evaluates the feasibility of laparoscopic surgery in patients diagnosed with colorectal liver metastases. Half of participants will be operated on by laparoscopic approach and the results obtained will be compared with the results from the other half of patients operated on by open approach.

DETAILED DESCRIPTION:
The safety and efficacy of liver surgery in the treatment of colorectal liver metastases are well established for the open approach. It allows good results in terms of complications, disease free survival and overall survival, and for these reasons it has become the gold standard technique in the treatment of colorectal liver metastases.

On the contrary, the role of laparoscopic liver resection in this context is not so clear nowadays. Generally, laparoscopic surgery offers some advantages such as less pain, shorter hospital stay and better aesthetic results. But the use of laparoscopic approach in liver surgery is still discussing: two international consensus conferences have been held and no strong conclusions have been made. Furthermore for colorectal liver metastases no randomized trials, comparing both techniques, have been published until now.

To assess the feasibility of laparoscopic liver resection for colorectal metastases, the investigators propose this trial in which the patients suitable for laparoscopic approach are randomized to open or laparoscopic group

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal liver metastases;
* Patients suitable for surgical treatment;
* Patients eligible for laparoscopy approach.

Exclusion Criteria:

* Patients with high tumour load: multiples and bilobar colorectal metastases;
* Patients with big liver metastases or close to major vessels;
* Patients with oncological contraindications for surgery;
* Cirrhotic liver
* Needing for two stage liver resection;
* Medical or psychiatric condition of the patient that compromises the informed consent authorization;
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

SECONDARY OUTCOMES:
Surgical operative time | Intraoperative
  Duration of the surgical intervention
Blood losses | Intraoperative
  Blood loss in milliliter
Transfusion | Intraoperative
  Number of blood transfusions required during surgical operation
Hospital stay | Up to 3 months
  Days between surgical operation and hospital discharge
Time between surgery and adjuvant chemotherapy | Up to 3 months
  Days between surgical operation and the beginning of adjuvant chemotherapy
Mortality | 90 days
Morbidity | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Robles Campos, MD; PHD, Study Chair — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Universitario "Virgen de la Arrixaca", Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robles-Campos R, Lopez-Lopez V, Brusadin R, Lopez-Conesa A, Gil-Vazquez PJ, Navarro-Barrios A, Parrilla P. Open versus minimally invasive liver surgery for colorectal liver metastases (LapOpHuva): a prospective randomized controlled trial. Surg Endosc. 2019 Dec;33(12):3926-3936. doi: 10.1007/s00464-019-06679-0. Epub 2019 Jan 30. PMID 30701365